CLINICAL TRIAL: NCT03465202
Title: A Prospective Evaluation of Capecitabine and Metabolite Pharmacokinetics in Elderly Breast and Colorectal Cancer Patients and Their Association With Toxicity and Molecular Markers of Enzyme Activity and Aging
Brief Title: Association of Capecitabine Pharmacokinetics and Toxicity With Aging
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: University of Newcastle Upon-Tyne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SBRU201501
Record Dates: First submitted 2015-08-07; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: Capecitabine; Pharmacokinetics; Ageing; Frailty; Breast cancer; Colorectal cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Frailty | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine (Experimental)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
This is a multi-centre prospective non-interventional study designed to evaluate the effects of patient age on the pharmacokinetics of capecitabine and its metabolites 5'DFCR, 5'DFUR, and 5-FU. In addition, the study will assess the correlation between the pharmacokinetic parameters calculated and cytidine deaminase, biomarkers of aging, clinical frailty, treatment outcome, and toxicity. To be enrolled, patients must have breast or colorectal cancer and be eligible to receive capecitabine monotherapy in accordance with its approved clinical usage in the UK. Treatment will be administered according to NICE guidelines as well as the clinical judgement of the prescribing physician. One hundred patients (50 breast cancer patients, 50 colorectal cancer patients) who are about to start treatment with capecitabine monotherapy will be recruited to the study and undergo study procedures within the first week of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Histologic or cytologic diagnosis of breast cancer or colorectal cancer. Patients should have disease that is suitable for capecitabine monotherapy as defined by the NICE Guidelines.

  2) Patients must be within the first week of their first cycle of capecitabine treatment.

  3) Estimated life expectancy of greater than 3 months. 4) Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2. 5) Total serum bilirubin less than or equal to 25 micromol/L. 6) Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than 2.5 times the upper limit of the normal range.

  7) Serum albumin level greater than 32 g/L. 8) Creatinine clearance greater than or equal to 30 mL/minute. 9) Blood haemoglobin level of greater than 9 g/dL, with transfusion allowed. 10) Absolute neutrophil count greater than 2.5 x 109/L. 11) Platelet count greater than 100 x 109/L. 12) 18 years of age or older. 13) Written informed consent.

Exclusion Criteria:

1. Pregnancy or breast feeding.
2. Known HIV, Hepatitis B, or Hepatitis C infection.
3. Known Gilbert syndrome.
4. Uncontrolled diabetes (HbA1c greater than 7.5%).
5. Any condition or disease that might affect oral absorption of medications, including:

   1. Crohn's disease
   2. Ulcerative colitis
   3. Major gastric or small bowel resection

      -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of capecitabine and metabolites | 0 (pre-dose), 0.5, 1, 2, 4, and 6 hours post dose
  Measurement of AUC of capecitabine and its metabolites 5'deoxy-5-fluorocytidine (5'DFCR), 5'deoxy-5-fluorouridine (5'DFUR), and 5-fluorouracil.

SECONDARY OUTCOMES:
Toxicities and grades as scaled by Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.03 | Six months
  Toxicity grade(s) as measured by CTCAE version 4.03 (published by the U.S. Department of Heath and Human Services 2009). General grading scheme is as follows: Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL). Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Progression free survival as measured by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 | From time of enrollment until first documented progression
  Progression free survival as measured by the RECIST criteria version 1.1 (Eisenhauer et al., 2009). The RECIST criteria define progression as 'at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: the appearance of one or more new lesions is also considered progression)'
Response as measured by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 | From time of enrollment to first documented response
  Complete or partial response as measured by the RECIST criteria version 1.1. (Eisenhauer et al., 2009) Complete response = 'Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial response = 'At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.'
Grip strength measured in kg | During 6-hour pharmacokinetic study session
  Grip strength measured in kg by the grip strength test (using the Takei handheld dynamometer)
Frailty as measured by the Edmonton Frail Scale | During 6-hour pharmacokinetic study session
  Frailty as measured by the Edmonton Frail Scale. A 17 point scale that measures 9 frailty domains. 0-5: not frail; 6-7: vulnerable; 8-9: mild frailty; 10-11: moderate frailty; 12-17: severe frailty.
Nutritional status as measured by the Mini Nutritional Assessment questionnaire | During 6-hour pharmacokinetic study session
  Nutritional status as measured by the Mini Nutritional Assessment questionnaire, a 30 point test on nutritional status. Scoring: 24 to 30 points: Normal nutritional status.
  17 to 23.5 points: At risk of malnutrition. Less than 17 points: malnourished.
Quality of life as assessed by the European Organization for Research and Treatment of Cancer quality of life (EORTC-QLQ-C30 version 3) questionnaire | During 6-hour pharmacokinetic study session
  Quality of life as measured by the EORTC-QLQ-C30 version 3 questionnaire. This questionnaire assesses the quality of life of cancer patients in a series of 30 questions, with 28 of the questions on a scale of 1 to 4 where 1 is 'not at all' and 4 is 'very much'. Final two questions relate to overall quality of life and health on a scale of 1 to 7, where 1 is 'very poor' and 7 is 'excellent'.
Plasma cytidine deaminase activity (measured in units/mg protein by spectrophotometric assay) | 0 hours post dose (pre-dose)
  Plasma cytidine deaminase activity (measured in units/mg protein by spectrophotometric assay).
Maximum plasma concentration (Cmax) of capecitabine and metabolites | 0 (pre-dose), 0.5, 1, 2, 4, and 6 hours post dose
  Cmax of capecitabine and its metabolites 5'deoxy-5-fluorocytidine (5'DFCR), 5'deoxy-5-fluorouridine (5'DFUR), and 5-fluorouracil.
Time of maximum plasma concentration (Tmax) of capecitabine and metabolites | 0 (pre-dose), 0.5, 1, 2, 4, and 6 hours post dose
  Cmax of capecitabine and its metabolites 5'deoxy-5-fluorocytidine (5'DFCR), 5'deoxy-5-fluorouridine (5'DFUR), and 5-fluorouracil.